CLINICAL TRIAL: NCT03141541
Title: Does a Patient Education Focused on Pain Management Improve Disability, Pain Coping and Quality of Life in Patients With Low Back Pain and Psychosocial Risk Factors?
Brief Title: Pain Management for Patients With Low Back Pain and Psychosocial Risk Factors in a Hospital Setting.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6300005
Record Dates: First submitted 2017-03-03; First posted 2017-05-05 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain
Keywords: low back pain; cognitive behavioural therapy; randomised controlled trial
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Parallel group randomised controlled trial
Who Masked: Investigator
Masking Description: The invistigator performing the data analysis is unaware of group allocation. Due to the study design (pain management intervention versus usual care) it is not possible to blind patients and care providers.
  Furthermore, as outcomes are selfreported, masking of assessors is not possible, as the patients are the assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): All patients receive a thorough physical examination by a rheumatologist or a chiropractor with a subsequent examination by a physiotherapist.The patients receive general information about the nature back pain, adjustment of analgesic treatment and clarification of any need of further diagnosing or assessment by a surgeon. The physiotherapist furthermore makes an assessment of the patients' physical capacity and function and provides guidelines for any exercise programme. Based on the physiotherapist's judgement, the patient may be referred to rehabilitation in the local community
- Group based pain management intervention (Experimental): In addition to usual care as described for the control group, the patients in the intervention group will participate in a cognitive group-based pain management intervention. The aim of the intervention is to improve the patients' understanding of their back pain problem, and that they learn different pain coping strategies. The intervention is based on cognitive behavioural therapy including elements of acceptance and commitment therapy, and furthermore uses different relaxation and breathing exercises.
  Interventions: Behavioral: Group based pain management intervention

INTERVENTIONS:
Behavioral: Group based pain management intervention — The intervention is delivered as six separate sessions of each two hours duration over a four month period. The sessions are managed by a multidisciplinary team from the Spine Center, led by a psychologist. Before the first session, each patient in the intervention group participates in an individual consultation with the psychologist or nurse, with the aim of matching expectations for the group intervention, and hereby ensure the patients compliance throughout the intervention.
  Arms: Group based pain management intervention

SUMMARY:
Patients with low back pain and coexisting psychosocial risk factors have a poorer prognosis in terms of quality of life, disability, sick leave and health care use. Despite existing literature showing that low back pain patients benefit from cognitive therapy interventions, this has not been investigated in subgroups of low back pain patients with psychosocial risk factors.

The purpose of the study is to investigate whether patients referred to secondary care with low back pain and coexisting psychosocial risk factors will have a better treatment outcome when participating in a pain management course in addition to usual care.

This will be investigated in a randomised study design, where 130 patients with chronic low back pain and psychosocial risk factors will be randomly allocated to either usual care or a cognitive-therapy based pain management intervention in addition to usual care.

The patients will be followed for one year after inclusion, and patientreported outcomes on disability, pain, sick leave, quality of life and pain coping will be collected by the use of questionnaires at baseline, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-specifick low back pain lasting ≥ 3 months
* Psychosocial risk profile defined as a fear avoidance score >24 (Örebro Musculoskeletal Pain Questionnaire) and/or a bodily distress score >15 (Common Mental Disorder Questionnaire) and/or health anxiety score >9 (Common Mental Disorder Questionnaire)
* Speaks and understands Danish
* Age ≥ 18 years

Exclusion Criteria:

* Inflammatory or malignant disease
* Spine surgery within the last year
* Untreated or severe depression
* Psychiatric course of treatment within the last year
* Abuse of drugs or alcohol
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire | Change from baseline to 12 months after baseline
  The Roland-Morris is a 24-item self-report questionnaire about how low-back pain affects functional activities. Each question is worth one point so scores can range from 0 (no disability) to 24 (severe disability).

SECONDARY OUTCOMES:
Low Back Pain Rating Scale - Back pain | Change from baseline to 12 months after baseline
  In the present study only the pain index of the LBPRS is used. The LBPRS pain index consists of two subscales, which measure back pain and leg pain, respectively. On each subscale the intensity of back pain and leg pain are reported on a 0-10 scale (best-worst) using the following three questions: the pain intensity at the time of examination, the average pain intensity within the past two weeks and the worst pain experienced within the past two weeks. The score of each subscale are reported separately (0-10 scale).
Low Back Pain Rating Scale - Leg pain | Change from baseline to 12 months after baseline
  In the present study only the pain index of the LBPRS is used. The LBPRS pain index consists of two subscales, which measure back pain and leg pain, respectively. On each subscale the intensity of back pain and leg pain are reported on a 0-10 scale (best-worst) using the following three questions: the pain intensity at the time of examination, the average pain intensity within the past two weeks and the worst pain experienced within the past two weeks. The score of each subscale are reported separately (0-10 scale).
EuroQol 5 Dimensions | Change from baseline to 12 months after baseline
  The EQ-5D is a measure of generic quality of life. It comprises five dimensions, which are mobility, selfcare, usual activities, pain/discomfort and anxiety/depression. Each dimension has three levels (no problem, some problems, extreme problems) resulting in a total of 245 potential health states. The scores fall on a scale of -0.624 to 1.000 (perfect health) including the scores of -0.293 for "unconscious" and 0.000 for "dead".
Pain Catastrophizing Scale | Change from baseline to 12 months after baseline
  The PCS measures an individual's pain experience through 13 questions asking about how one feels and what he/she thinks about when in pain. The PCS evaluates pain catastrophizing as a single construct with three components: rumination, magnification, and helplessness. Each question is answered on a 0-4 scale (best worst), adding up to a total score of 0-52 (best-worst).
Sick leave | Change from baseline to 12 months after baseline
  The patients report their average weekly sick leave during the past 4 weeks in the three categories 0 days per week, 1-4 days per week, 5-7 days per week, all the time.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Rolving, PhD, Principal Investigator — Diagnostic Centre, Silkeborg Regional Hospital
Locations (1):
- Diagnostic Centre, Regional Hospital Silkeborg, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The data will be available to other researchers when the study results have been published (anticipated 2020). The data will be available on request from the authors.